CLINICAL TRIAL: NCT00355615
Title: A Phase IIIb, Efficacy, and Safety Study of Rosuvastatin in Children 10-17 Years of Age With Heterozygous Familial Hypercholesterolemia: a 12-week, Double-blind, Randomized, Multicenter, Placebo-controlled Study With a 40-week, Open-label, Follow-up
Brief Title: PLUTO: Pediatric Lipid-redUction Trial of rOsuvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3561C00087; PLUTO
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Results first posted 2009-07-20 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Familial Hypercholesterolemia
Keywords: Heterozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Rosuvastatin Calcium; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- rosuva 5 (Active Comparator): rosuvastatin 5 mg
  Interventions: Drug: Rosuvastatin
- rosuva 10 (Active Comparator): rosuvastatin 10 mg
  Interventions: Drug: Rosuvastatin
- rosuva 20 (Active Comparator): rosuvastatin 20 mg
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- rosuva ol (Other): rosuvastatin open label
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — oral
  Other Names: Nexium
  Arms: rosuva 10; rosuva 20; rosuva 5; rosuva ol
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of once-daily rosuvastatin in reducing LDL-C in children and adolescents aged 10-17 years with HeFH from baseline (Day 0) to the end of the 12-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (at least 1 year post-menarche) children and adolescents (aged 10 -17 years) with heterozygous familial hypercholesterolemia (HeFH)

Exclusion Criteria:

* Certain medical conditions and lab test results
* History of a reaction to rosuvastatin or other statin drugs
* Use of specified disallowed medications

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crestor Medical Science Director, MD, Study Director — AstraZeneca
Locations (20):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, Hyde Park, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Wexford, Pennsylvania
- Canada (5):
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Sherbrook, Quebec
- Netherlands (7):
  - Research SIte, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Hoorn
  - Research Site, Rotterdam
  - Research Site, Utrecht
  - Research SIte, Waalwijk
- Research Site, Oslo, Norway
- Spain (3):
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Reus

REFERENCES:
- [Derived] Avis HJ, Hutten BA, Gagne C, Langslet G, McCrindle BW, Wiegman A, Hsia J, Kastelein JJ, Stein EA. Efficacy and safety of rosuvastatin therapy for children with familial hypercholesterolemia. J Am Coll Cardiol. 2010 Mar 16;55(11):1121-6. doi: 10.1016/j.jacc.2009.10.042. PMID 20223367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred male and female (Tanner stages II to V, at least 1 year post-menarche) children and adolescents (aged 10 to 17 years with Heterozygous familial hypercholesterolemia were randomized into the study, from 20 sites located in The United States (3 sites), The Netherlands (7 sites), Norway (1 site), Spain (3 sites), and Canada (6 sites).
Pre-assignment Details: Patients entered a 6 week dietary lead-in/drug washout period. Eligible patients were then randomly assigned to double-blind treatment with rosuvastatin 5 mg, 10 mg, 20 mg, or matching placebo, administered orally once daily for 12 weeks.
Period: Randomized Double Blind Period
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo | Rosuva ol
Started | 42 | 44 | 45 | 46 | 0 (open label phase followed the randomized phase)
Completed | 41 (1 dropped out due to adverse event) | 44 | 44 (45 were randomized but 1 never received drug) | 45 (1 dropped out due to an adverse event) | 0
Not Completed | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0
Period: 40-week Rosuvastatin Open Label Period
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo | Rosuva ol
Started | 0 | 0 | 0 | 0 | 173
Completed | 0 | 0 | 0 | 0 | 164
Not Completed | 0 | 0 | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3
Not completed — investigational site closed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo | Total
Number analyzed (Participants) | 42 | 44 | 45 | 46 | 177
Age Continuous [Mean (Full Range); unit: years] | 14.1 [10 to 17] | 14.5 [11 to 17] | 14.2 [11 to 17] | 14.3 [10 to 17] | 14.3 [10 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 22 | 24 | 97
  Male | 16 | 19 | 23 | 22 | 80
Baseline low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 237.70 (55.06) | 229.10 (44.70) | 237.40 (47.80) | 229.00 (43.13) | 233.3 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline (Day 0) to the End of the 12-week Double-blind Treatment Phase
Description: Percent change in low-density lipoprotein cholesterol (LDL-C) = (final value - Baseline value)/Baseline value * 100
Time Frame: 12 weeks
Population: Intention-to-treat (ITT) analysis set included all randomized patients who took study medication and had both a baseline reading and at least 1 post-baseline reading for the variable being analyzed. Analyses were performed using the last-observation-carried-forward (LOCF) method on the ITT analysis set for all efficacy outcome variables.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
percentage | -38.5 (11.38) | -44.4 (12.15) | -50.2 (13.3) | -0.5 (13.18)

2. Secondary Outcome: Percent Change in LDL-C and Other Lipid Parameters From Baseline to Week 6, and at End of Double-blind Dose Treatment Phase (Week 12)
Description: Percent change from baseline in LDL-C after six week of treatment
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
percentage | -40.3 (12.22) | -45.2 (11.15) | -50.0 (11.42) | -0.6 (13.63)

3. Secondary Outcome: Percent Control Rate Based on Achievement of LDL-C Target of <110 mg/dL During Double-blind Dose Treatment
Description: Percent of patients achieving LDL-C < 110 mg/dL out of the total patients in each treatment group
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
Percent of Participants | 11.9 | 40.9 | 40.9 | 0.0

4. Secondary Outcome: Percent Change in HDL-C
Description: Percent change in high-density lipoprotein cholesterol (HDL-C) after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
percent change | 4.5 (15.53) | 10.1 (14.19) | 8.9 (14.11) | 7.6 (17.89)

5. Secondary Outcome: Percent Change in Non-HDL-C at 12 Weeks
Description: Percent change in non-HDL-C at 12 weeks
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
percent change | -36.3 (9.98) | -42.8 (11.50) | -47.7 (13.50) | -0.8 (11.89)

6. Secondary Outcome: Percent Change in Triglycerides (TG)
Description: Percent change in tryglycerides (TG) after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
percent change | 2.6 (49.07) | -14.2 (29.66) | -7.9 (55.88) | 3.4 (48.27)

7. Secondary Outcome: Percent Change in Total Cholesterol (TC)
Description: Percent change from baseline in total cholesteral after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
percent change | -30.0 (9.63) | -34.1 (9.5) | -38.9 (12.08) | 0.2 (10.53)

8. Secondary Outcome: Percent Change in Apolipoprotein A-1 (ApoA-1)
Description: Percent change in ApoA-1 after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 43 | 43 | 46
mean percent change | 2.3 (9.69) | 4.3 (9.85) | 3.9 (10.68) | 3.6 (15.59)

9. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB)
Description: Percent change in ApoB after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 43 | 43 | 46
mean percent change | -32.1 (9.13) | -37.8 (11.75) | -40.7 (13.91) | -1.5 (14.67)

10. Secondary Outcome: Percent Change in ApoB/ApoA-1
Description: Percent change in the ratio of ApoB/ApoA-1 after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 43 | 43 | 46
mean percent change | -33.1 (9.99) | -40.0 (12.06) | -42.8 (12.23) | -3.4 (16.70)

11. Secondary Outcome: Percent Change in LDL-C/HDL-C
Description: Percent change in the ratio of LDL-C/HDL-C after 12 weeks of treatment
Time Frame: After 12 week of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
mean percent change | -40.4 (11.36) | -48.6 (13.26) | -53.6 (12.85) | -5.5 (17.98)

12. Secondary Outcome: Percent Change in TC/HDL-C
Description: Percent change in the ratio of TC/HDL-C after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
mean percent change | -32.1 (10.72) | -39.3 (11.55) | -43.2 (11.76) | -5.2 (15.03)

13. Secondary Outcome: Percent Change in Non-HDL-C/HDL-C
Description: Percent change in the ratio of non-HDL-C/HDL-C after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo
Number analyzed (Participants) | 42 | 44 | 44 | 46
mean percent change | -37.9 (12.12) | -47.1 (13.12) | -51.2 (13.18) | -5.8 (17.63)

ADVERSE EVENTS:
Arm/Group | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo | Rosuva ol
Serious Adverse Events (participants affected / at risk) | 0 | 0 | 0 | 1 | 2
Other Adverse Events (participants affected / at risk) | 12 | 14 | 17 | 17 | 75
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo | Rosuva ol
Appendicitis (Infections and infestations) | 0/42 | 0/44 | 0/44 | 0/46 | 1/173
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0/42 | 0/44 | 0/44 | 0/46 | 1/173
Vision Blurred (Eye disorders) | 0/42 | 0/44 | 0/44 | 1/46 | 0/173
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Rosuva 5 | Rosuva 10 | Rosuva 20 | Placebo | Rosuva ol
Fatigue (General disorders) | 1/42 | 1/44 | 1/44 | 0/46 | 9/173
Headache (Nervous system disorders) | 6/42 | 7/44 | 9/44 | 9/46 | 29/173
Influenza (Infections and infestations) | 2/42 | 2/44 | 0/44 | 4/46 | 14/173
Nasopharyngitis (Infections and infestations) | 3/42 | 7/44 | 7/44 | 5/46 | 36/173
Nausea (Gastrointestinal disorders) | 2/42 | 0/44 | 2/44 | 2/46 | 10/173
Tonsillitis (Gastrointestinal disorders) | 0/42 | 0/44 | 3/44 | 1/46 | 2/173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less